CLINICAL TRIAL: NCT05496790
Title: Role of Lipoprotein(a) in Patients With Cardiovascular Diseases and Young Patients With Premature Acute Coronary Syndromes
Brief Title: Role of LipoprotEin(a) in CardiovascuLar Diseases and Premature Acute Coronary Syndromes - (RELACS) Study
Acronym: RELACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Arturo Cesaro, Assistant Professor, University of Campania Luigi Vanvitelli
Other Study IDs: CECN/1385
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Acute Coronary Syndrome; Lipoprotein Disorder; Acute Myocardial Infarction; Cardiovascular Diseases
Keywords: Lipoprotein(a); Lp(a); Acute Coronary Syndrome (ACS); Acute Myocardial Infarction; Premature ACS
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several clinical and preclinical studies have focused interest on lipoprotein(a) [Lp(a)], showing a direct and independent relationship of its circulating levels with the progression of atherosclerosis and its clinical manifestations. However, to date, Lp(a) represents an underestimated predictor of CV risk, especially in higher-risk populations, such as patients with strong CV familiarity and recurrent and/or early-onset CV events.

The key point of the project will be the evaluation of the role of Lp(a) in the development of atherosclerotic disease and, specifically, acute coronary syndrome.

DETAILED DESCRIPTION:
Although acute myocardial infarction (AMI) is more common in the elderly, its incidence in young patients is increasing. The exact pathogenetic mechanism of AMI in young patients remains largely unknown and involves the interaction of multiple genetic and environmental factors related to atherothrombosis. The cardiovascular risk profile and coronary artery disease burden differ between young and elderly patients with AMI. Generally, compared with elderly patients, patients with premature AMI have a lower atherosclerotic burden, as well as a lower incidence of hypertension and diabetes mellitus. Still, they more frequently have a hypercoagulable state with high fibrinogen and D-dimer levels and genetic disorders of lipid metabolism (1) with elevated triglyceride and lipoprotein (a) [Lp(a)] levels (2).

Lp(a) is a lipoprotein with pro-atherogenic, pro-thrombotic and pro-inflammatory properties (3). Lp(a) consists of a lipid component with apoB100 and a protein component represented by Apo(a)(3,4). Apo(a) shows substantial structural homology with plasminogen, suggesting that the former protein can inhibit the binding of plasminogen to its receptor, thereby interfering with fibrinolysis and inducing a prothrombotic state. Several studies have shown that increased plasma levels of Lp(a) are associated with an increased risk of coronary artery disease (5), peripheral arteriopathy (6), cerebrovascular disease (7), abdominal aortic aneurysm, aortic valve stenosis and calcification (8), and venous thromboembolism (9). In addition, elevated Lp(a) levels are associated with an increased risk of major cardiac adverse events (10). In contrast, a recent study that included approximately 1,500 patients with a history of acute coronary syndrome (ACS) at least six months after enrollment showed that Lp(a) appears to be an independent risk factor for ACS in individuals <45 years young (especially in the presence of LDL-C cholesterol levels >70 mg/dL) (11). This association is of lesser magnitude (but still preserved) between 45-60 years of age and becomes nonsignificant after 60 years of age. Despite increasing evidence in the literature, Lp(a) determination is infrequently performed in patients with early-onset ACS referred to Cardiology Departments and Outpatient Departments. Therefore, hyper-Lp(a) remains largely under-diagnosed even in patients at high or very high cardiovascular risk.

Therefore, the purpose of our study is to evaluate the correlation between Lp(a) and recurrence of cardiovascular events such as cardiovascular mortality, recurrence of anginal symptoms, new revascularizations (PCI/CABG), or new hospitalizations at 1-year follow-up in patients with premature ACS, which includes myocardial infarction with ST-segment elevation (STEMI), acute myocardial infarction without ST-segment elevation (NSTEMI) and unstable angina (UA).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Documented coronary artery disease (i.e.,acute coronary syndrome [ACS], percutaneous coronary intervention [PCI], coronary artery bypass graft surgery [CABG], and at least one of the following:

  1. at least one CV event before 60 years of age;
  2. multiple CV events despite optimal medical therapy.
* Signature of informed consent.

Exclusion Criteria:

* Age > 60 years
* Patients experiencing cardiogenic shock and unable to provide informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18-60 years with documented coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Impact of Lp(a) on MACE | Through study completion, an average of 1 year
  Assess at a 1-year follow-up, the impact of Lp(a) on the major cardiovascular events (MACE) defined as cardiovascular mortality, recurrence of anginal symptoms, new revascularizations (PCI/CABG), stroke, or new hospitalizations for cardiovascular causes.

SECONDARY OUTCOMES:
Each component of the primary enpoint | Through study completion, an average of 1 year
  To assess the incidence of cardiovascular events individually such as cardiovascular mortality, recurrence of anginal symptoms, new revascularizations (PCI/CABG), stroke, or new hospitalizations for cardiovascular causes at 1-year follow-up, in patients with elevated Lp(a) levels.
Lp(a) levels in premature ACS | Through study completion, an average of 1 year
  To assess Lp(a) levels in subjects with early-onset acute coronary syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- AORN S. Anna e S. Sebastiano, Caserta, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cesaro A, Schiavo A, Moscarella E, Coletta S, Conte M, Gragnano F, Fimiani F, Monda E, Caiazza M, Limongelli G, D'Erasmo L, Riccio C, Arca M, Calabro P. Lipoprotein(a): a genetic marker for cardiovascular disease and target for emerging therapies. J Cardiovasc Med (Hagerstown). 2021 Mar 1;22(3):151-161. doi: 10.2459/JCM.0000000000001077. PMID 32858625
- [Background] Gragnano F, Fimiani F, Di Maio M, Cesaro A, Limongelli G, Cattano D, Calabro P. Impact of lipoprotein(a) levels on recurrent cardiovascular events in patients with premature coronary artery disease. Intern Emerg Med. 2019 Jun;14(4):621-625. doi: 10.1007/s11739-019-02082-8. Epub 2019 Mar 30. No abstract available. PMID 30929131